CLINICAL TRIAL: NCT03931421
Title: B Cell Maturation Antigen（BMCA）-Targeted CAR-T for Refractory/Relapsed Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Wenbin Qian, clinical professor, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lymphoma center Q004
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: In this trial, T cells were seperated from refractory/relapsed multiple myeloma patients and engineered into BMCA-targeted CAR-T cells, and then transfused back into the patients for the treatment of their multiple myeloma.
Masking Description: It's an open-label trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experiment group (Experimental): In this arm, patients are treated with B Cell Maturation Antigen (BMCA)-targeted CAR-T cells and the safety and efficacy will be observed.
  Interventions: Biological: CAR-T treatment

INTERVENTIONS:
Biological: CAR-T treatment — a novel method for treatment of multiple myeloma, in which patients' T cells are engineered into B Cell Maturation Antigen（BMCA）-Targeted CAR-T cells to eliminate myeloma cells.

SUMMARY:
It's a single arm, open label prospective study, in which the safety and efficacy of B Cell Maturation Antigen（BMCA）-targeted CAR-T thearpy are evaluated in refractory/relapsed multiple myeloma patients.

DETAILED DESCRIPTION:
In this trial, T cells are seperated from multiple myeloma patients, and engineered into BMCA-targeted CAR-T cells, these cells are then transfused back into the patients to elimimnate the myeloma cells. In this process, the safety and efficacy of this CAR-T treatment are closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age≥18，male or female;
* 2. ECOG 0-3;
* 3. Clearly diagnosed as multiple myeloma (MM) [according to IMWG 2014 criteria];
* 4. Patients should have received 3 different regimens prior to enrollment (each regimen should last for at least one complete cycle, except for the case of disease progression);
* 5. Previously received one PI and IMiD treatment;
* 6. MM patients should fit one of the following: 1) disease progression; 2) relapsed after CR. The corresponding criteria is defined as follows: a, disease progression should satisfy at least 1 of the following: serum M protein ≥0.5g/dl, or urine M protein>200mg/24h, or FLC increasement >10mg/dl, or bone marrow plasma cell proportion >10%, or with new bone disease/plasmacytoma/original focus increased by 50% or more, or hypercalcemia ( corrected serum calcium level >11.5mg/dL(2.65mmol/L); b. relapse after CR, should satisfy one of the following: ①M protein in urine or blood; ②bone marrow plasma cell proportion≥5%; ③manifestation of disease progression, such as plasmacytoma, osteolytic lesions or hypercalcemia.
* 7. Peripheral blood mononucleated cell separation should be at least 2 weeks from chemo/radiotherapy;
* 8. Neutrophil count≥1000/ul, platelet count≥45000/ul, Hb>60g/l;
* 9. Cardiac, hepatic and renal function: Creatinin <1.5 times of normal maximum；ALT/AST level <2.5 times of the maximum of normal range; total bilirubin<1.5 times of ULN；cardiac ejection fraction≥ 50%; no pericardial effusion within 6 weeks prior to enrollment;
* 10. Being able to understand and willing to sign the written consent;
* 11. Fertile patients should agree to take contraceptive measures during the process of this trial.

Exclusion Criteria:

* 1. History of other tumors other than multiple myeloma, except for the following: malignant tumor after radical surgery, and have been inactive for ≥3 years prior to enrollment; skin cancer (not melanoma) after sufficient treatment, no evidence of disease at enrollment;
* 2. History of the following treatment: received targeted therapy, epigenetic therapy or clinical trials, invasive operation within 14 days/5 half-time prior to enrollment. History of monoclonal antibody within 21 days prior to enrollment. History of cytotoxic medicine or proteasome treatment within 14 days prior to enrollment. History of immunomodulatory treatment within 7 days prior to enrollment;
* 3. History of >5mg/d systemic prednisone treatment (or other glucocorticoids of the equivalent dosage) within 2 weeks prior to peripheral mononucleated cell collection;
* 4. With CNS involvement or clinical manifestation of meningeal myeloma;
* 5. With active systemic infection;
* 6. With active HBV infection or HCV infection, or history of type C hepatitis;
* 7. With immunodeficiency, including HIV infection;
* 8. With the following heart condition: NYHA level III or IV congestive heart failure; myocardial infarction or CABG within 6 months prior to enrollment; clinically meaningful ventricular arrythmia, or history of idiopathic syncope (not caused by vascular-vagal disorder or dehydration), history of non-ischemic myopathy;
* 9. With active autoimmune disease;
* 10. History of autologous stem cell transplantation within 6 weeks prior to enrollment;
* 11. History of allogenic stem cell transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-31 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | at the time point 3 months after CAR-T cell transfusion
  complete remission rate after treated by CAR-T therapy
incidence and severity of adverse events | from the date of the start of treatment to 36 months after last patient's enrollment
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure

SECONDARY OUTCOMES:
progression free survival | from the day of treatment to the date of first documented progression，up to 36 months after the last patient's enrollment
  from date of inclusion to date of progression, relapse, or death from any cause
overall survival | from the day of treatment to the date of first documented progression，up to 36 months after the last patient's enrollment
  from the date of inclusion to date of death, irrespective of cause
duration of the CAR-T cells in the patients | from the date of re-transfusison to 36 months after last patient's enrollment
  time from re-transfusion to date when the modified T cells become non-detectable

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
All the data would be available on the website of the affiliated hospital after the trial is completed
Supporting Information: Study Protocol, CSR